CLINICAL TRIAL: NCT01477164
Title: Effects of Aerobic and Resistance Training on Accumulation of Old, Modified Proteins in Young and Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K. Sreekumaran Nair, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-005853
Record Dates: First submitted 2011-09-28; First posted 2011-11-22 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Sarcopenia
Keywords: Exercise; Aging; Sarcopenia; Muscle function
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aerobic Exercise Training (Experimental): Participants will perform 12-weeks of high intensity aerobic training.
  Interventions: Behavioral: High intensity aerobic exercise
- Combined (Active Comparator): The combined group will have 12-weeks of no exercise followed by 12-weeks of combined aerobic and resistance exercise training. Assessments will be made at three time points: baseline, after 12-weeks of no training, and after 12-weeks of combined training.
  Interventions: Behavioral: Combined
- Resistance Exercise Training (Experimental): Participants will perform 12-weeks of resistance exercise training.
  Interventions: Behavioral: Resistance exercise training

INTERVENTIONS:
Behavioral: High intensity aerobic exercise — Participants will perform 12-weeks of high intensity aerobic training. Training will be 5-days per week. Three days (e.g. Monday, Wednesday and Friday) will include repeated bouts of cycling for 4-minutes at ~90% maximal effort followed by 3 minutes of active rest. The other two days (e.g. Tuesday and Thursday) will be treadmill exercise for 45 minutes at 70% of maximal effort.
  Arms: Aerobic Exercise Training
Behavioral: Resistance exercise training — Participants will perform 12-weeks of resistance exercise training. Training will be 5-days per week of daily sessions of 60 minutes that include resistance exercise for all major muscle groups.
  Arms: Resistance Exercise Training
Behavioral: Combined — The combined group will be assessed before and after 12 weeks of no exercise training, then again following 12 weeks of combined aerobic and resistance exercise training.
  Arms: Combined

SUMMARY:
Muscle proteins accumulate damage during aging and leads to the loss of muscle mass and function in older people. Exercise can increase the making of new proteins and removal of older proteins, but it is not known if the effect changes with aging or type of exercise. The investigators will determine the ability for endurance, resistance, or a combination of exercise training to remove older-damaged proteins and make newer-functional muscle proteins in groups of younger and older people. The investigators will particularly study protein that are involved with energy production (mitochondrial proteins) and force production (contractile proteins).

Hypothesis 1: Older people will have greater accumulation of damaged proteins than younger people.

Hypothesis 2: Aerobic exercise will decrease the accumulation of damaged forms of contractile and mitochondrial proteins in younger and older people.

Hypothesis 3: Resistance exercise will decrease the accumulation of damaged forms of contractile proteins in younger and older people.

DETAILED DESCRIPTION:
The loss of muscle mass and function with age leads to high social and economic costs. Lifestyle interventions that can help maintain muscle mass and function can be beneficial to improve health and decrease the costs associated with loss of independence in the elderly. Muscle proteins accumulate damage during aging, which is suggested to lead to loss of function. The biological processes that remove damaged proteins and synthesis new proteins appear to be decreased with aging. Exercise is known to increase the processes that remove older and synthesis newer muscle proteins and may be an effect lifestyle intervention to improve muscle quality and function. Additionally, specific types of proteins appear to decay with age including contractile and mitochondrial proteins. Different types of exercise training can increase the making of specific proteins. The investigators will examine the ability for aerobic and resistance training to increase the quality of mitochondrial and contractile proteins between younger and older people.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* 18 to 30 years or 65 to 80 years old
* Male and female

Exclusion Criteria:

* Regular exercise program
* Smoking
* Metabolic disease (diabetes, cardiovascular disease, cancer, thyroid disorders)
* Pregnancy
* Inability to exercise
* Overweight or obesity
* Drugs known to impair metabolic function (statin, beta-blocker, anti-inflammatory)
* Allergies to lidocaine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-11; Primary Completion 2016-05 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle protein synthesis rate | Approximately 14 weeks for the endurance or resistance training groups and approximately 28 weeks for the combined group
  The investigators will determine the rate of incorporation of stable isotope amino acid tracers in skeletal muscle proteins during several hours of rest. The measurement will be an average resting muscle protein synthesis rate (% new muscle protein per hour) and will be performed at baseline and following 12 weeks of exercise training.

CONTACTS AND LOCATIONS:
Overall Officials: K. Sreekumaran Nair, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Pataky MW, Heppelmann CJ, Sevits KJ, Asokan AK, Kumar AP, Klaus KA, Dasari S, Kunz HE, Strub MD, Robinson MM, Coon JJ, Lanza IR, Adams CM, Nair KS. Aerobic and resistance exercise-regulated phosphoproteome and acetylproteome modifications in human skeletal muscle. Nat Commun. 2025 Jul 1;16(1):5700. doi: 10.1038/s41467-025-60049-0. PMID 40595512
- [Derived] Zhang X, Habiballa L, Aversa Z, Ng YE, Sakamoto AE, Englund DA, Pearsall VM, White TA, Robinson MM, Rivas DA, Dasari S, Hruby AJ, Lagnado AB, Jachim SK, Granic A, Sayer AA, Jurk D, Lanza IR, Khosla S, Fielding RA, Nair KS, Schafer MJ, Passos JF, LeBrasseur NK. Characterization of cellular senescence in aging skeletal muscle. Nat Aging. 2022 Jul;2(7):601-615. doi: 10.1038/s43587-022-00250-8. Epub 2022 Jul 15. PMID 36147777